CLINICAL TRIAL: NCT03572049
Title: SUBA-itraconazole Versus Conventional Itraconazole in the Treatment of Endemic Mycoses: a Multi-center, Open-label Comparative Trial
Brief Title: Endemic Mycoses Treatment With SUBA-itraconazole vs Itraconazole
Acronym: MSG15
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, Davis (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Peter Pappas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSG15; MSG-15 (Other: Mycoses Study Group); UTN U1111-1228-5154 (Other: World Health Organization)
Record Dates: First submitted 2018-02-01; First posted 2018-06-28 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-09

CONDITIONS: Invasive Fungal Infections
Keywords: Histoplasmosis; Coccidioidomycosis; Blastomycosis
MeSH Terms: conditions — Invasive Fungal Infections; Histoplasmosis; Coccidioidomycosis; Blastomycosis | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUBA itraconazole (Experimental): Stage 1: Day 1-3 two 65 mg capsules three times daily with food. Days 4-42 two 65 mg capsules twice daily with food.
  Stage 2 : Days 43-180 two 65 mg capsules twice daily with food
  Interventions: Drug: SUBA itraconazole
- Conventional itraconazole (Active Comparator): Stage 1: Day 1-3 two 100 mg capsules three times daily with food. Days 4-42 two 100 mg capsules twice daily with food.
  Stage 2 : Days 43-180 two 100 mg capsules twice daily with food
  Interventions: Drug: Conventional itraconazole

INTERVENTIONS:
Drug: SUBA itraconazole — SUBA itraconazole study drug will consist of two 65 mg capsules to be taken three times a day with food for days 1-3 of study. For days 4-180 of study, two 65mg capsules will be taken twice daily with food.
  Arms: SUBA itraconazole
Drug: Conventional itraconazole — Conventional itraconazole comparator drug will consist of two 100 mg capsules to be taken three times a day with food for days 1-3 of study. For days 4-180 of study, two 100 mg capsules will be taken twice daily with food.
  Other Names: itraconazole; Sporanox
  Arms: Conventional itraconazole

SUMMARY:
This is a prospective, multi-center, randomized, open-label parallel arm study involving patients with proven or probable invasive endemic fungal infection to ascertain the pharmacokinetics, safety, efficacy, tolerability and health economics of oral SUBA-itraconazole compared to conventional itraconazole. Patients will receive randomized open-label study drug (SUBA-itraconazole or conventional itraconazole) over a 42 day period and then continue therapy until Day 180. Patients will be stratified based on clinically reported infection with the human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, open-label parallel arm study involving patients with proven or probable invasive endemic fungal infection to ascertain the pharmacokinetics, safety, efficacy, and tolerability of oral SUBA-itraconazole or itraconazole. Patients will receive randomized open-label study drug (either SUBA- itraconazole 130 mg twice daily or itraconazole 200 mg twice daily) over a 42-day period and then continue on their assigned open-label therapy until day 180.

The study sample size will be 80 evaluable patients - target enrollment (three arms: approximately 40 histoplasmosis, 20 coccidioidomycosis, 20 other endemic fungal infections).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age > 18 years who have given written informed consent to participate
2. Patients with a proven or probable endemic mycosis (Histoplasma, Coccidioides, Paracoccidioides, Blastomyces, Sporothrix, Talaromyces marneffei (formerly Penicillium marneffei) according to current EORTC/MSG (Mycoses Study Group) criteria, including patients who:

   * Are immunosuppressed, including as a result of HIV/AIDS
   * Have had a heart, lung or bone marrow transplant
   * Have had chemotherapy for cancer
   * Are otherwise normal hosts

Exclusion Criteria:

1. Significant liver dysfunction as evidenced by at least 5 times greater than upper limits of normal baseline ALT (alanine aminotransferase) , AST (aspartate aminotransferase), alkaline phosphatase, or total bilirubin.
2. Use of an alternative antifungal therapy (IV or oral) for more than 14 days for this infection, with the exception of Coccidioidomycosis. Subjects with Coccidioidomycosis who previously received fluconazole therapy for more than 14 days may be included, if in the opinion of the investigator, they are having an inadequate response or, are intolerant of fluconazole (e.g. due to adverse events). Such subjects must washout from fluconazole for 7 days (~5 half-lives of fluconazole) before starting investigational therapy.
3. Evidence of CNS (central nervous system) infection.
4. Unable to take PO medications.
5. Female patients who are lactating or pregnant.

   Women should be:
   1. Postmenopausal for 1 year,
   2. Post-hysterectomy or bilateral oophorectomy,
   3. If of child bearing potential have a negative β-HCG (human chorionic gonadotropin) at screening and using highly effective method of birth control throughout course of study or remain abstinent for duration of study.
6. Documented intolerance, allergy or hypersensitivity to an azole.
7. Inability to comply with study treatment, study visits, and study procedures.
8. Known history of congestive cardiac failure on medical treatment, fungal endocarditis, or other causes of ventricular dysfunction that may outweigh the benefit of itraconazole.
9. Patients with active TB (tuberculosis)
10. Concurrent use of astemizole, rifampin/rifampicin, rifabutin, ergot alkaloids, long acting barbiturates, carbamazepine, pimozide, quinidine, neostigmine, terfenadine, ketoconazole, valproic acid, or St. John's wort in the 5 days prior to first administration of study drug.
11. Any known or suspected condition of the patient that may jeopardize adherence to the protocol requirements or impede the accurate measurement of efficacy.
12. Treatment with any investigational agent in the 30 days prior to study entry.
13. Patients unlikely to survive 30 days (including severe fungal disease defined by systolic blood pressure (SBP) < 90; hypoxia < 60).
14. Patients with body weight < 40 kg.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Pappas, MD, Principal Investigator — University of Alabama at Birmingham; George R Thompson, MD, Study Chair — University of California, Davis; Andrej Spec, MD, Principal Investigator — Washington University School of Medicine
Locations (12):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California at Davis, Sacramento, California
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Metro Infectious Disease Associates, Overland Park, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Unniversity of Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin, Madison, Wisconsin
- Hospital Santo Tomás, Panama City, Panama

REFERENCES:
- [Derived] Spec A, Thompson GR, Miceli MH, Hayes J, Proia L, McKinsey D, Arauz AB, Mullane K, Young JA, McGwin G, McMullen R, Plumley T, Moore MK, McDowell LA, Jones C, Pappas PG. MSG-15: Super-Bioavailability Itraconazole Versus Conventional Itraconazole in the Treatment of Endemic Mycoses-A Multicenter, Open-Label, Randomized Comparative Trial. Open Forum Infect Dis. 2024 Jan 29;11(3):ofae010. doi: 10.1093/ofid/ofae010. eCollection 2024 Mar. PMID 38440302
- [Derived] Thompson GR 3rd, Lewis P, Mudge S, Patterson TF, Burnett BP. Open-Label Crossover Oral Bioequivalence Pharmacokinetics Comparison for a 3-Day Loading Dose Regimen and 15-Day Steady-State Administration of SUBA-Itraconazole and Conventional Itraconazole Capsules in Healthy Adults. Antimicrob Agents Chemother. 2020 Jul 22;64(8):e00400-20. doi: 10.1128/AAC.00400-20. Print 2020 Jul 22. PMID 32457106

RESULTS

PARTICIPANT FLOW:
Groups:
- SUBA Itraconazole: Stage 1: Day 1-3 two 65 mg capsules three times daily with food. Days 4-42 two 65 mg capsules twice daily with food.
  Stage 2 : Days 43-180 two 65 mg capsules twice daily with food
  SUBA itraconazole: SUBA itraconazole study drug will consist of two 65 mg capsules to be taken three times a day with food for days 1-3 of study. For days 4-180 of study, two 65mg capsules will be taken twice daily with food.
- Conventional Itraconazole: Stage 1: Day 1-3 two 100 mg capsules three times daily with food. Days 4-42 two 100 mg capsules twice daily with food.
  Stage 2 : Days 43-180 two 100 mg capsules twice daily with food
  Conventional itraconazole: Conventional itraconazole comparator drug will consist of two 100 mg capsules to be taken three times a day with food for days 1-3 of study. For days 4-180 of study, two 100 mg capsules will be taken twice daily with food.
Period: Overall Study
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Started | 42 | 46
Completed | 33 | 35
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUBA Itraconazole | Conventional Itraconazole | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Continuous [Mean (Full Range); unit: years] | 53 [18 to 79] | 48 [19 to 80] | 50 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 27 | 32 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Plasma Itraconazole Levels and Hydroxyitraconazole Levels at Day 14
Description: Percentage of participants to achieve therapeutic itraconazole and hydroxyitraconazole levels by evaluating Inter-patient variability as calculated by co-efficient of variation on plasma specimens collected on Day 14
Time Frame: Day 14
Measure: Number; unit: percentage of participants
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Number analyzed (Participants) | 42 | 46
percentage of participants | 60.5 | 71.0

2. Primary Outcome: Frequency of Treatment Related Adverse Events Days 1-42
Description: Comparison of the number of treatment related adverse events in each arm occurring Days 1-42.
Time Frame: Day 42
Measure: Number; unit: adverse events
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Number analyzed (Participants) | 42 | 46
adverse events | 15 | 27

3. Secondary Outcome: Comparison of Plasma Itraconazole Levels and Hydroxyitraconazole Levels at Day 42
Description: Percentage of patients with therapeutic itraconazole and hydroxyitraconazole levels as measured in plasma trough levels Day 42
Time Frame: Day 42
Measure: Number; unit: percentage of participants
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Number analyzed (Participants) | 42 | 46
percentage of participants | 69.3 | 58.0

4. Secondary Outcome: Resolution of Signs and Symptoms of Invasive Fungal Infection on Day 42
Description: We will measure specific signs and symptoms related to endemic fungal infection, comparing baseline findings to Day 42 findings using physical examination and patient history.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Number analyzed (Participants) | 37 | 40
Participants | 29 | 30

5. Secondary Outcome: The Number of Days of Hospitalization at Day 180
Description: The number of days of Hospitalization occurring between Day 1-180
Time Frame: Day 180
Measure: Mean (Full Range); unit: Days
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
Number analyzed (Participants) | 42 | 46
Days | 5 [0 to 50] | 7 [0 to 50]

ADVERSE EVENTS:
Time Frame: Data regarding all adverse events were collected over 180 days (approximately 6 months).
Arm/Group | SUBA Itraconazole | Conventional Itraconazole
All-Cause Mortality (participants affected / at risk) | 1/42 | 0/46
Serious Adverse Events (participants affected / at risk) | 4/42 | 12/46
Other Adverse Events (participants affected / at risk) | 16/42 | 22/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUBA Itraconazole (N=42) | Conventional Itraconazole (N=46)
UTI Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypomolar Nonketotic Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Edema, lower extremities (Vascular disorders) | 1 (1) | 1 (1)
Hypertrophic Obstructive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Pain in foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (3)
Liver Toxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ascites, worsening (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Motor Vehicle Accident (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Gastro-intestinal hemorrhage with hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea, worsening (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea, worsening (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Catheterization (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUBA Itraconazole (N=42) | Conventional Itraconazole (N=46)
Weight Gain (General disorders) | 2 (3) | 0 (0)
Weakness (General disorders) | 4 (4) | 0 (0)
Rash (General disorders) | 3 (3) | 4 (4)
Pruritus (General disorders) | 3 (3) | 0 (0)
Night sweats (General disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (7)
Lightheadedness (General disorders) | 2 (2) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Insomnia (Nervous system disorders) | 3 (3) | 0 (0)
Hypertension (Cardiac disorders) | 4 (4) | 8 (8)
Headache (Nervous system disorders) | 4 (5) | 7 (7)
Fever (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 4 (4) | 0 (0)
Emesis (Gastrointestinal disorders) | 2 (2) | 7 (7)
Edema (Cardiac disorders) | 12 (17) | 10 (12)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 10 (11)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (5)
Blurry Vision (General disorders) | 2 (2) | 0 (0)
Anorexia (General disorders) | 3 (4) | 0 (0)
Weight loss (General disorders) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dyspnea (Reproductive system and breast disorders) | 0 (0) | 4 (5)
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Chest Pain (Cardiac disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03572049/Prot_SAP_001.pdf